CLINICAL TRIAL: NCT03489213
Title: NExT (Nutrition and Exercise Cancer Survivor Trial)
Brief Title: Nutrition and Exercise Trial: Improving Diet and Physical Activity Patterns in Overweight Cancer Survivors
Acronym: NExT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Steven Clinton, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OSU-17012; NCI-2017-01031 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2018-02-09; First posted 2018-04-05 (Actual); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Cancer Survivor; Overweight
MeSH Terms: conditions — Overweight | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (DGA/AICR) (Active Comparator): Patients receive DGA/AICR-based dietary intervention for 6 months consisting of 12 education sessions (60 minutes each) every other week. Lectures will take place in an urban garden where fruit, vegetable, and herb harvesting 1-2 times per week is encouraged. All participants will be given a FitBit and regular physical activity will be encouraged. Finally, remote health coaching is offered to all study subjects for the duration of the intervention (12 weeks).
  Interventions: Other: Dietary Intervention; Behavioral: Exercise Intervention; Other: Laboratory Biomarker Analysis; Dietary Supplement: Nutritional Intervention; Other: Questionnaire Administration
- Arm II (DGA/AICR plus Beef) (Experimental): Patients receive the same intervention as in Arm I with the addition of 18 ounces of lean beef provided by the study to each subject. Subjects will be encouraged to consume the lean beef and lectures will incorporate healthy beef consumption into each lesson and cooking demonstration.
  Interventions: Other: Dietary Intervention; Behavioral: Exercise Intervention; Other: Laboratory Biomarker Analysis; Dietary Supplement: Nutritional Intervention; Other: Questionnaire Administration

INTERVENTIONS:
Other: Dietary Intervention — Participants randomized to the DGA/AICR group will receive plant-based diet education, garden access and health coaching for 5 months. The sessions are offered every other week.
  Other Names: Dietary Modification; intervention, dietary; Nutrition Intervention; Nutrition Interventions; Nutritional Interventions
Behavioral: Exercise Intervention — Participants will wear a FitBit every day and monitor daily physical activity.
Other: Laboratory Biomarker Analysis — Correlative studies
Dietary Supplement: Nutritional Intervention — Participants randomized to the beef group will receive 11 to 18 ounces of frozen lean beef each week for home preparation, in addition to DGA/AICR diet education, garden access and health coaching.
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized phase II trial will enroll overweight cancer survivors. Subjects in both groups will be educated to follow a diet pattern similar to what is recommended by the Dietary Guidelines for Americans and the American Institute for Cancer Research (DGA/AICR) but one group will also receive 18 ounces of lean beef for incorporation into a healthy diet. Subjects will be encouraged to exercise regularly and activity will be monitored throughout the study. Nutrition and exercise may help cancer survivors successfully maintain improved dietary patterns, body composition, and physical activity efforts and consumption of beef may favorably impact lean body mass and specific nutritional outcomes.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility and compliance with a the Dietary Guidelines for Americans/American Institute for Cancer Research (DGA/AICR) healthy dietary pattern and a beef + DGA/AICR healthy dietary pattern in cancer survivors.

II. To determine the impact of dietary interventions on body composition, clinical outcomes, and physical performance.

III. To quantify the impact of the two dietary interventions on cardiometabolic biomarkers of health.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive DGA/AICR-based dietary intervention for 6 months consisting of 12 education sessions over 60 minutes every other week, fruit, vegetable, and herb harvesting 1-2 times per week for 2 hours, wearing a FitBit during physical activity, and remote health coaching over 10 minutes for 12 weeks.

ARM II: Patients receive DGA/AICR-based dietary intervention as in Arm I and consume 11-18 ounces of lean beef each week for 6 months.

Clinical and physical activity assessments will take place at baseline, after the intervention and at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index (BMI) >= 25 kg/m^2
* Be non-vegetarian/non-vegan, and have no concerns with beef consumption
* Have completed active curative therapy for cancer within the past 36 months (i.e., surgery, chemotherapy, or radiation); ongoing hormone therapy is acceptable
* Voluntarily provide consent, Health Insurance Portability and Accountability Act (HIPPA) authorization form, and consent from primary care provider (PCP) or treating oncologist
* Not be planning to travel for more than 3 consecutive weeks during the intervention period
* Agree to refrain from all nutritional supplements, herbal supplements, and botanical supplements aside from those prescribed by a physician for the duration of the study

Exclusion Criteria:

* Are cognitively unable to consent or have physical or mental limitations that would prevent full participation in the program
* Are vegan or those unwilling to consume 11-18 ounces (oz) of beef per week
* Have pre-existing medical conditions that preclude unsupervised physical activity (i.e., severe orthopedic conditions, impending hip or knee replacement, paralysis, unstable angina, dementia, recent history of myocardial infarction, congestive heart failure, pulmonary conditions requiring oxygen, or hospitalization in past 6 months)
* Have had cancer treatment that significantly impacts digestion, metabolism, or food intake (e.g., surgical loss of esophagus, stomach, or colon, pancreas dysfunction, or brain surgery that alters cognition, etc.)
* Report meeting the recommendations for physical activity (> 60 minutes per day, most days per week) and already meet the majority of dietary guidelines as assessed by a telephone screener
* Are prescribed medication that do not allow for increased intake of fruits and vegetables
* Have recently (< 3 months) started a statin or other lipid lowering medication; participants who report that they are changing a lipid lowering drug dose or drug type during the recruitment period will also be excluded; participants who have been stable on a lipid-lowering medication for at least 3 months may participate; well-controlled diabetics (type I or II) may participate
* Have been diagnosed with active metabolic or digestive illnesses (i.e., Celiac disease, irritable bowel syndrome [IBS], renal insufficiency, hepatic insufficiency)
* Are pregnant or are planning to become pregnant during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2017-04-25 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Adherence to either the DGA/AICR group or the DGA/AICR + Beef group | Up to 12 months
  Participants will keep both 7 day diet records periodically through out the study as well as a daily log of beef consumption
Change in body composition | Up to 12 months
  Change in body composition will be assessed by dual X-ray absorptiometry (iDXA)
Change in blood pressure | Baseline up to 12 months
  Trained personnel will use a sphygomanometer to assess blood pressure
Change in body mass index (BMI) | Baseline up to 12 months
  Weight and height will be combined to report BMI in kg/m^2.
Change in dietary carotenoid intake | Baseline up to 12 months
  Assessed by Raman spectroscopy
Change in blood carotenoids | Up to 12 months
  Assessed by High Pressure Liquid Chromatography
Change in physical performance assessed by timed performance-related mobility tasks | Baseline up to 12 months
  Physical performance will be measured using the 40 M walk test
Change in physical performance | Up to 12 months
  Assessed by a standardized stair climb test
Dietary intake patterns | Up to 6 months
  Will be assessed using diet logs maintained throughout the intervention and graphical food frequency questionnaire (FFQ). This FFQ automatically calculates the Healthy Eating Index 2010. Will use previous 30-day intake for all FFQs to assess dietary patterns. To determine protein balance, will use a 7-day diet record prior to a 24-hr urine collection.
Adherence to classes | Up to 12 months
  Descriptive statistics will be generated using attendance forms
Change in fasting glucose | Up to 12 months
  A fasting blood sample will be used to measure glucose at three time points
Change in lipoprotein profiles | Up to 12 months
  A fasting blood sample will be used to assess serum lipoprotein profile
Daily physical activity (steps per day) | up to 12 months
  Each participants daily FitBit data will be downloaded to a secure spreadsheet

SECONDARY OUTCOMES:
Health related quality of life | Up to 12 months
  Measured at all three time points using the Health Related Quality of Life (HR-QOL) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Steven Clinton, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- [Derived] Hill EB, Pashkova A, Grainger EM, Roberts KM, Chitchumroonchokchai C, Braun AC, Ralston RA, Riedl KM, Spees CK, Clinton SK. Targeted Urinary Profiling as a Biomarker of Dietary Flavonoid Intake from Fruits and Vegetables and its Relationship to the Timing of Dietary Assessment. Curr Dev Nutr. 2025 Jul 31;9(9):107520. doi: 10.1016/j.cdnut.2025.107520. eCollection 2025 Sep. PMID 41080470
- [Derived] Braun AC, Portner J, Grainger EM, Clinton SK, Xu M, Darragh A, Pratt KJ, Weaver LL, Spees CK. Impact of Dietitian-Delivered Motivational Interviewing Within a Food is Medicine Intervention Targeting Adults Living With and Beyond Cancer. J Cancer Educ. 2025 Aug;40(4):609-615. doi: 10.1007/s13187-024-02552-4. Epub 2024 Dec 21. PMID 39708224
- See also: The Jamesline — http://cancer.osu.edu